CLINICAL TRIAL: NCT03056651
Title: Day-care Unit for Patients With Refractory Heart Failure - a Single-centre Study
Brief Title: Day-care Unit for Patients With Refractory Heart Failure
Acronym: DayCare-HF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Silesian Centre for Heart Diseases (Other)
Responsible Party: Principal Investigator, Mariusz Gasior, MD, PhD, Professor, Silesian Centre for Heart Diseases
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DayCare-HF; DCHFU (Other: Silesian Centre for Heart Disease)
Record Dates: First submitted 2017-02-12; First posted 2017-02-17 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Heart Failure; Heart Diseases; Cardiovascular Diseases
Keywords: heart failure; day care; prognosis
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DayCare-HF (Other): Comprehensive service in day-care unit, including education, diagnostic tools (i.e. electrocardiography, transthoracic echocardiography, implanted cardioverter defibrillator (ICD) / cardiac resynchronization therapy device (CRT) interrogation and possibility of intravenous drug administration (i.e. loop diuretics, dobutamine).
  Interventions: Other: treatment in day-care heart failure unit

INTERVENTIONS:
Other: treatment in day-care heart failure unit

SUMMARY:
The Day-Care Unit for Patients With Refractory Heart Failure (DayCare-HF) is an observational study on selected patients with advanced refractory heart failure. The purpose of the study was to examine the comprehensive management of HF in the day-care unit in terms of the safety and its impact on the rehospitalization and mortality rates in patients with advanced refractory HF.

DETAILED DESCRIPTION:
The Day-Care Unit for Patients With Refractory Heart Failure (DayCare-HF) is a single-center observational study conducted in the 3rd Department of Cardiology, School of Medicine with the Division of Dentistry in Zabrze, Medical University of Silesia in Katowice, Silesian Centre for Heart Disease in Zabrze, Poland.

The main objective of the DayCare-HF is to verify the hypothesis that comprehensive and multidisciplinary day-care management of patients with refractory heart failure (HF) is safe and beneficial in terms of hospital readmission due to HF and al cause mortality.

The study population is formed by selected patients with heart failure, hospitalized in cardiology wards and intensive cardiac care unit of Silesian Centre for Heart Disease, who fulfilled eligibility criteria.

During the scheduled visits comprehensive medical service is provided, including education, diagnostic tools (electrocardiography, transthoracic echocardiography, implanted cardioverter defibrillator (ICD) / cardiac resynchronization therapy device (CRT) interrogation and additional treatment (intravenous loop diuretic, dobutamine, vasodilators administration).

The patients are under constant follow-up for major adverse events, heart transplantation, hospital readmissions due to HF and all cause mortality.

ELIGIBILITY:
Inclusion Criteria:

1. Optimally decongested heart failure in New York Heart Association (NYHA) class II-IV, treated for at least 6 months
2. Performance of all possible reparative procedures if indications were present (cardiac revascularization, correction of valvular heart disease, cardiac ablation, cardiac resynchronization therapy)
3. Implantation of cardioverter-defibrillator (ICD) if applicable
4. At least two unplanned hospitalizations for heart failure during preceding 6 months

Exclusion Criteria:

1. Inability to travel to the unit
2. Non-compliance with the medical recommendations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with rehospitalization due to heart failure decompensation | From date of inclusion until the date of death from any cause, assessed up to 1 year

SECONDARY OUTCOMES:
Number of participants with major adverse cardiovascular event | From date of inclusion until the date of death from any cause, assessed up to 1 year
Number of participants with reported deaths from any cause | From date of inclusion until the date of death from any cause, assessed up to 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Silesian Centre for Heart Disease, Zabrze, Silesian Voivodeship, Poland